CLINICAL TRIAL: NCT06624995
Title: Comparison of Traditional Nurse-led Education and Chatbot on the Prevention of Postoperative Complications After Major Visceral Surgery: a Randomized Controlled Trial
Brief Title: Chatbot on the Prevention of Postoperative Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer at medical surgical nursing, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0637
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Visceral Surgery Complications

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditional nurse-led education (No Intervention)
- chatbot education (Experimental)
  Interventions: Other: chatbot education

INTERVENTIONS:
Other: chatbot education — elderly patients interacted with Chatbot to discuss general postoperative complication related inquiries
  Arms: chatbot education

SUMMARY:
Major visceral surgery encompasses a broad range of operations with a wide variety of procedures that fall under this category. The majority of patients undergoing major visceral surgery often present with cancer and other medical comorbidities and are put at an elevated risk of a large number of medical and surgical postoperative complications

DETAILED DESCRIPTION:
Complications following major visceral surgery are relatively common and are estimated to occur in 18-23% of patients . The management of complications is challenging for both the elderly patient and the perioperative team, and adds considerably to the cost of care particularly when further interventions involve readmission, unplanned admission to an intensive care unit, interventional radiology and/or an unplanned return to theatre. With the advancement of online patient portals, the use of internet to seek for health information is already a common phenomenon; Chatbot may become a more significant source of information for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years old and above, both sex, scheduled for elective major visceral surgery, able to communicate in the local language, and without any cognitive impairment.

Exclusion Criteria:

* Elderly patients with a history of major psychiatric disorders, patients with a history of previous major visceral surgery, and patients who were unable to provide informed consent will be excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
postoperative morbidity | patient will be evaluated at three time points: 24 hour postoperative; 48 hours postoperative , and 30 days postoperative.
  using the postoperative morbidity survey , Patients are assessed for diagnostic features in nine domains (pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, haematological, wound and pain). For each of the nine domains morbidity is recorded on the presence or absence of preset criteria and it appears to accurately describe the pattern and prevalence of morbidity in the postoperative setting. I

SECONDARY OUTCOMES:
Geriatric anxiety | will be measured at three time points: 90 to 120 minutes before the preoperative consultation (baseline ); after 7 days postoperative, and after 30 days postoperative
  questionnaire comprising 30 items, called the GAS was created to evaluate, screen for, and quantify the intensity of anxiety symptoms in older persons
quality of life | will be measured at two time points : at baseline (preoperative ) and after 30 days postoperative
  This short version of the SF-36 tool consists of 12 items and eight scales: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and perceived mental health (MH).
usability of using chatbots | 4 weeks postoperatively
  This scale was composed of 16 validated items aimed to assess the personality, onboarding, navigation, understanding, responses, error handling and intelligence of a chatbot.

IPD SHARING:
Plan to Share IPD: No